CLINICAL TRIAL: NCT04563403
Title: Improving the Efficacy of Exposure Therapy Using Projection-Based Augmented Reality for the Treatment of Cockroach Phobia: A Randomized Clinical Trial
Brief Title: Improving the Efficacy of Exposure Therapy for the Treatment of Cockroach Phobia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Jaume I (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TERA-P MS SS
Record Dates: First submitted 2020-09-21; First posted 2020-09-24 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Specific Phobia, Animal
Keywords: Specific Phobia; Cockroach phobia; Exposure therapy; Projection-Based augmented reality therapy; Multiple Stimuli; Single Stimulus; Randomized Clinical Trial
MeSH Terms: conditions — Phobia, Specific

STUDY DESIGN:
Intervention Model Description: Randomized Clinical Trial with two treatment conditions
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment with Multiple Stimuli (Experimental): Projection-based augmented reality therapy (P-ARET) with Multiple Stimuli (MS) (P-ARET MS). Intervention group that receives P-ARET treatment varying the stimuli available in the system (different cockroaches in colour, size, etc).
  Interventions: Behavioral: Projection-based augmented reality therapy (P-ARET)
- Treatment with Single Stimuli (Experimental): Projection-based augmented reality therapy (P-ARET) with Single Stimuli (SS) (P-ARET SS). Intervention group that receives P-ARET treatment using a single stimulus (one cockroach).
  Interventions: Behavioral: Projection-based augmented reality therapy (P-ARET)

INTERVENTIONS:
Behavioral: Projection-based augmented reality therapy (P-ARET) — The intervention will be based on exposure therapy to cockroaches using P-ARET. The treatment will follow the guidelines of the "one-session treatment" (OST). Main components: Psychoeducation, Exposure to the feared object (cockroach), modeling (the therapist will interact with the phobic stimulus first and if possible, the patient will follow the same steps), cognitive challenge, and reinforcement and relapse prevention.

SUMMARY:
The aim of this study is to test the efficacy and efficiency of the Projection-Based augmented reality therapy under two conditions: multiple stimuli (different types of cockroaches) (P-ARET MS) versus single stimulus (one cockroach) (P-ARET SS) for the treatment of participants diagnosed with cockroach phobia.

DETAILED DESCRIPTION:
Specific phobia (SP) refers to an extreme and persistent fear of a specific object or situation that is out of proportion to the actual danger or threat. SP is the most prevalent anxiety disorder with substantial impairment and comorbidity. Animal fear is one of the most prevalent subtypes of SP. In vivo exposure is the treatment of choice for this problem, but this technique presents limitations in its implementation related to the access and acceptability (i.e., low acceptance on the part of patients and therapists, high dropout rates, limited access to the treatment and, difficulties in its application in the clinical context). Augmented Reality (AR) offers some advantages in delivering the exposure technique: 1) Exposure to multiple virtual stimuli; 2) Going beyond reality; 3) Allowing complete control over the situation; 4) It allows privacy and confidentiality. Particularly, the most significant aspect of AR is that the virtual elements add relevant and helpful information to the physical information available in the real world.

We pretend to go a step beyond and explore ways of optimizing exposure therapy based on the inhibitory learning approach. AR can maximize some strategies like "variability" (varying stimuli, durations, levels of intensity, or the order of the hierarchy items), greater control by the therapists or "exposure to multiple contexts" which can produce a positive effect in terms of fear renewal and generalization of the results. Therefore, the aim of this study is to test the efficacy and efficiency of varying the phobic stimuli during the ARET: using multiple stimuli (MS) (P-ARET MS) versus single stimulus (SS) (P-ARET SS) in participants with cockroach phobia.

The Randomized Clinical Trial (RCT) will be conducted following the Consolidated Standards of Reporting Trials (CONSORT: http://www.consort-statement.org) and the SPIRIT guidelines (Standard Protocol Items: Recommendations for Intervention Trials). Participants (N = 80) who received a diagnosis of SP for cockroaches (DSM-5), will be randomized into two experimental conditions: 1) Projection-based augmented reality therapy (P-ARET) with Multiple Stimuli (MS) (P-ARET MS); 2) Projection-based augmented reality therapy (P-ARET) with Single Stimulus (SS) (P-ARET SS). Five evaluation moments will be included: pre-intervention, post- intervention, and 1-, 6- and 12-month follow-ups.

ELIGIBILITY:
Inclusion Criteria:

* Being at least 18 years old
* Meeting DSM-5 diagnostic criteria for SP (animal subtype) to cockroaches -
* Having a minimum of six-month duration of the phobia
* Sign an informed consent
* Presenting a score of at least 4 on the fear and avoidance scales of the diagnostic interview applied

Exclusion Criteria:

* Presence of another severe mental disorder that requires immediate attention
* Having current alcohol or drug dependence or abuse, psychosis or severe organic illness
* Currently being treated in a similar treatment program
* Being capable of inserting their hands in a plastic container with a cockroach (during the behavioral test)
* Receiving other psychological treatment during the study for cockroach phobia
* Start receiving pharmacological treatment during the study (or in case of being already taking them, change the drug or dose)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-11-30 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in Behavioral Avoidance Test (BAT; adapted from Öst, Salkovskis, & Hellström's, 1991). | Baseline ( At the beginning of the intervention) and immediately after the intervention, and at 1, 6 and 12 months after the end of the treatment.
  Patients will be confronted to a real cockroach and they will be encouraged to get closer and interact with the stimulus as much as they can. The anxiety level (0-10), distance and level of interaction with the animal will be registered and evaluated in a scale ranging from 0 (the participant does not enter the room) to 12 (the participant interacts with the cockroach).

SECONDARY OUTCOMES:
Change in Behavioral Avoidance Test through AR (BAT; adapted from Öst, Salkovskis, & Hellström's, 1991). | Baseline ( At the beginning of the intervention) and immediately after the intervention, and at 1, 6 and 12 months after the end of the treatment.
  Patients will be confronted to a novel projected cockroach (not used before in any of the two treatment conditions) and they will be encouraged to get closer and interact with the stimulus as much as they can. The anxiety level (0-10), distance and level of interaction with the animal will be registered and evaluated in a scale ranging from 0 (the participant does not enter the room) to 12 (the participant interacts with the cockroach).
Change in Fear of Cockroaches Questionnaire (adapted from Fear of Spiders Questionnaire; FSQ, Szymanski & O'Donohue, 1995). | Baseline ( At the beginning of the intervention) and immediately after the intervention, and at 1, 6 and 12 months after the end of the treatment.
  This questionnaire assesses the level of fear to cockroaches. It has 18 items evaluated in a scale ranging from 0 ("I strongly disagree") to 7 ("I strongly agree") ).
Change in Cockroach Phobia Beliefs Questionnaire (SBQ; adapted from Spider Phobia Beliefs Questionnaire; SBQ, Arntz, Lavy, van der Berg & van Rijssoort, 1993). | Baseline ( At the beginning of the intervention) and immediately after the intervention, and at 1, 6 and 12 months after the end of the treatment.
  This questionnaire assesses two different constructs, namely catastrophic beliefs about cockroaches and beliefs about the patient's own ability to cope with a cockroach. It has 78 items evaluated in a scale ranging from 0 (I don´t believe so) to 100 (I´m convinced of it).
Change in Fear and Avoidance Scales (adapted from Marks & Mathews, 1979). | Baseline ( At the beginning of the intervention) and immediately after the intervention, and at 1, 6 and 12 months after the end of the treatment.
  This instrument assesses the level of fear and avoidance to the feared stimulus (i. e., cockroaches), ranged from 0 (nothing) to 10 (very much). It evaluates target behavior, negative thoughts and modulators.
Change in Patient's Improvement Scale (adapted from the Clinical Global Impression scale; CGI, Guy, 1976). | Baseline ( At the beginning of the intervention) and immediately after the intervention, and at 1, 6 and 12 months after the end of the treatment.
  This instrument evaluates the degree of improvement of the patient's symptoms after the treatment compared to the start. It is ranged from 1 (much worse) and 7 (much better).
Change in Beck Depression Inventory 2nd edition (BDI-II; Beck, Steer, Brown, 1996; Spanish validation from Sanz, Navarro y Vázquez, 2003) | Baseline (At the beginning of the intervention) and immediately after the intervention, also at follow-up assessment periods (1, 6 and 12 months)
  This instrument assesses the existence and severity of symptoms of depression following the DSM-IV criteria. The BDI-II is a self report instrument that contains 21 items ranged from 0 to 3
Change in State-Trait Anxiety Inventory (adapted from Laux, Glanzmann, Schaffner, & Spielberger, 1981) | Baseline (At the beginning of the intervention) and immediately after the intervention, also at follow-up assessment periods (1, 6 and 12 months).
  This instrument includes two scales designed to assess state and trait anxiety respectively. Each scale contains 20 items ranged from 0 (nothing/rarely) to 3 (very much/always).

OTHER OUTCOMES:
Change in Anxiety Disorders Interview Schedule for DSM-IV-TR (ADIS-IV) | Baseline ( At the beginning of the intervention) and immediately after the intervention, and at 1, 6 and 12 months after the end of the treatment.
  Specific Phobia Diagnostic interview for specific phobia based on DSM-IV-TR criteria.
Change in Disgust Propensity and Sensitivity Scale-Revised-12 (DPSS-R-12; Sandín et al., 2008). | Baseline ( At the beginning of the intervention) and immediately after the intervention, and at 1, 6 and 12 months after the end of the treatment.
  This questionnaire includes two subscales that measure propensity to disgust and sensitivity to disgust. It contains 12 items ranged from 1 (never) to 5 (always).
Change in The Clinician Severity Scale (adapted from Di Nardo, Brown & Barlow, 1994). | Baseline ( At the beginning of the intervention) and immediately after the intervention, and at 1, 6 and 12 months after the end of the treatment.
  This instrument assesses the severity of symptoms evaluated by the clinician and the scale ranged from 0 (absent) to 8 (very severe).
Change in Scale of expectation and satisfaction with the treatment (adapted from Borkovec y Nau, 1972). | Baseline ( At the beginning of the intervention) and immediately after the intervention, and at 1, 6 and 12 months after the end of the treatment.
  This instrument contains 6 items ranged from 0 (nothing) to 10 (very much) assessing the patient's opinions about the treatment, focusing on their expectations and degree of satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- Universitat Jaume I, Castellon, Castellón, Spain

IPD SHARING:
Plan to Share IPD: Yes
According to the preservation of the privacy of the participants, the data from the clinical trial will be available upon reasonable request,
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Background] Shiban Y, Schelhorn I, Pauli P, Muhlberger A. Effect of combined multiple contexts and multiple stimuli exposure in spider phobia: A randomized clinical trial in virtual reality. Behav Res Ther. 2015 Aug;71:45-53. doi: 10.1016/j.brat.2015.05.014. Epub 2015 May 28. PMID 26072451
- [Background] Botella C, Mira A, Moragrega I, Garcia-Palacios A, Breton-Lopez J, Castilla D, Riera Lopez Del Amo A, Soler C, Molinari G, Quero S, Guillen-Botella V, Miralles I, Nebot S, Serrano B, Majoe D, Alcaniz M, Banos RM. An Internet-based program for depression using activity and physiological sensors: efficacy, expectations, satisfaction, and ease of use. Neuropsychiatr Dis Treat. 2016 Feb 23;12:393-406. doi: 10.2147/NDT.S93315. eCollection 2016. PMID 27042067
- [Derived] Palau-Batet M, Breton-Lopez J, Grimaldos J, Diaz-Sanahuja L, Quero S. Improving the efficacy of exposure therapy using projection-based augmented reality for the treatment of cockroach phobia: a randomised clinical trial protocol. BMJ Open. 2023 May 19;13(5):e069026. doi: 10.1136/bmjopen-2022-069026. PMID 37208142